CLINICAL TRIAL: NCT05044780
Title: Hyperspectral Analysis of Sweat Metabolite Biometrics for Real-Time Detection of COVID-19
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000178; 000178-C
Record Dates: First submitted 2021-09-14; First posted 2021-09-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: COVID-19
Keywords: camera; IL6; D-dimer; Coronavirus; SAR-COV-2; Natural History
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1/SARS-CoV-2 positive: Participants with molecular testing positive for SARS-CoV-2
- Cohort 2/SARS-CoV-2 negative: Participants with molecular testing negative for SARS-CoV-2

SUMMARY:
Background:

The COVID-19 pandemic has challenged the health systems worldwide. Many tools have been developed in response to the pandemic, but there is no current way to quickly screen multiple people for the disease. Research has shown that people with COVID-19 have higher levels of some proteins involved in the immune response and inflammation. These proteins can be detected in sweat using a special camera. Researchers want to see if analysis of sweat from fingerprints could be used to detect COVID-19 infection in people.

Objective:

To test a new technology to detect COVID-19 infection based on an analysis of sweat from fingerprints.

Eligibility:

Adults ages 18 and older who tested positive or negative for COVID-19 within the last 7 days.

Design:

Participants will visit the NIH Clinical Center for one day within 7 days from COVID-19 testing. The visit will last for 3 to 4 hours.

Participants who show symptoms for COVID-19 with a positive test will give blood samples to correlate with the sweat markers. About 1/2 tablespoon of blood will be drawn.

For sweat markers, 10 fingers will be imaged by a camera using a touchless system. This will be repeated 3 times. It will take about 15 minutes. Participants will use the device. They will get instructions and watch a short video on how to use the device.

DETAILED DESCRIPTION:
Background

The Coronavirus Disease 19 (COVID19) pandemic has challenged healthcare systems worldwide. Massive testing, contact tracing and social distancing proved to be the most effective tools to fight the pandemic prior to the development of vaccines.

Despite the effort to develop rapid diagnostic testing, we still don t have an available large population screening modality. Analysis of sweat metabolites from hyperspectral images of fingertips has the potential to be a valid clinic strategy to detect Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)infected individuals.

COVID19 has shown higher levels of inflammatory proteins like IL6, LDH, CRP, and d-dimer which have been implicated with severe COVID-19 induced pneumonitis and coagulopathy. These molecules can be detected as sweat metabolites and used as a biomarker for viral infection detection.

Objective

Identify a pattern classifier to distinguish between SARS-CoV-2 positive and SARS-CoV-2 negative human subjects by analysis of sweat metabolites from hyperspectral images of fingertips.

Eligibility

Individuals must all be >=18 years old

Must have standard of care molecular testing (either antigen or PCR) for SARS-CoV-2 within 7 days from study enrollment. Those individuals who tested positive will be enrolled in cohort 1 and those who tested negative will be enrolled in cohort 2

Study Design

This is an exploratory multisite study to evaluate the use of biometric analysis of sweat metabolites from hyperspectral images of fingertips to detect SARS-CoV-2 infection. Center for Cancer research (CCR), NCI will be the coordinating center.

All adult subjects that have available testing for SARS-CoV-2 completed within 7 days from the study enrollment are eligible for this study. The study will have two cohorts, cohort 1 (SARS-CoV-2 positive), and cohort 2 (SARS-CoV-2 negative). Fifty participants will be enrolled in each cohort to have hyperspectral imaging of the fingertips.

Every participant will have the right and left index fingers imaged by the camera with a touchless system. The imaging will be repeated three times. This imaging will take about 10 minutes.

The data obtained by the digital analysis will be compared to the result of the standard SARS-CoV-2 tests in use at the enrolling sites.

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligible subjects must meet the following inclusion criteria:

* Age >=18 years.
* Eligible for one of the following cohorts:

  * Cohort 1: Participants who tested positive for SARS-CoV-2 via standard of care molecular testing within 7 days of enrollment. Either antigen or PCR testing is acceptable. Results from home tests are not accepted.
  * Cohort 2: Participants must have a standard of care molecular testing negative for SARS-CoV-2 done within 7 days of enrollment. Either antigen or PCR testing is acceptable for enrollment. Results from home tests are not accepted.
* Ability of subject or Legally Authorized Representative (LAR) or Durable Power of Attorney (DPA) to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

Subjects with the following characteristics will be excluded from the study:

-Participants who have received remdesivir and/or dexamethasone for longer than 48 hours prior to hyperspectral imaging for the treatment of COVID19. Participants who have received up to 48 hours of treatment will be eligible.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will consist of two cohorts and each cohort will enroll 50 participants. Cohort 1 will enroll symptomatic participants who sought medical attention and tested positive for SARS-CoV-2, and Cohort 2 will enroll asymptomatic participants with a negative SARS-CoV-2 test.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Hyperspectal Analysis | One day
  Identify a pattern classifier to distinguish between SARS-CoV-2 positive (cohort 1) and SARS-CoV-2 negative (cohort 2) human subjects by hyperspectral analysis of sweat metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - INOVA Fairfax Medical Campus, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000178-C.html